CLINICAL TRIAL: NCT02972203
Title: MINDFUL-PC: Integrating Mindfulness Into the Patient-Centered Medical Home - A Pilot Study
Brief Title: MINDFUL-PC: Integrating Mindfulness Into the Patient-Centered Medical Home
Acronym: MINDFUL-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: The Arthur Vining Davis Foundations (Unknown); The Arnold P. Gold Foundation (Other)
Responsible Party: Principal Investigator, Zev Schuman Olivier, Research Director, Center for Mindfulness and Compassion, Cambridge Health Alliance
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB number: CHA-IRB-1002/08/14
Record Dates: First submitted 2016-11-04; First posted 2016-11-23 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Depression; Anxiety; Stress Related Disorder; Adjustment Disorder
Keywords: Mindfulness; primary care; self-control; self-regulation; adherence
MeSH Terms: conditions — Depression; Anxiety Disorders; Adjustment Disorders; Self-Control | interventions — Primary Health Care; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Training for Primary Care (Experimental): • Mindfulness Training for Primary Care (MPTC) is a primary care adaptation that includes core common Mindfulness-Based Intervention (MBI) elements. MTPC is a referral-based, insurance-reimbursable 8-week group psychotherapy delivered primarily by Patient-Centered Medical Home-integrated behavioral clinicians. MTPC groups are 2 hours long for 8 weeks, with a 7-hour day of silent group practice on a weekend. MTPC also emphasizes psychoeducational skills for self-regulation including a collaborative primary care provider (PCP) action-planning appointment during week 6.
  Interventions: Behavioral: Mindfulness Training for Primary Care
- Mindfulness Intro. +resources +waitlist (Active Comparator): Control arm: Participants receive a 60-minute introduction to mindfulness group plus referral to a list of community mindfulness resources such as private-pay community mindfulness classes, mobile mindfulness applications, books, and online recordings. These participants are added to a 6-month waitlist for a Cambridge Health Alliance (CHA) mindfulness-based intervention group. All participants are scheduled to meet with their primary care provider during week 6 for a collaborative action planning visit.
  Interventions: Behavioral: Mindfulness Intro. +resources +waitlist

INTERVENTIONS:
Behavioral: Mindfulness Training for Primary Care — • MPTC is a primary care adaptation that includes core common Mindfulness-Based Intervention (MBI) elements. MTPC is a referral-based, insurance-reimbursable 8-week group psychotherapy delivered primarily by Patient-Centered Medical Home-integrated behavioral clinicians. MTPC groups are 2 hours long for 8 weeks, with a 7-hour day of silent group practice on a weekend. MTPC also emphasizes psychoeducational skills for self-regulation including a collaborative primary care provider (PCP) action-planning appointment during week 6.
  Arms: Mindfulness Training for Primary Care
Behavioral: Mindfulness Intro. +resources +waitlist — Control arm: Participants receive a 60-minute introduction to mindfulness group plus referral to a list of community mindfulness resources such as private-pay community mindfulness classes, mobile mindfulness applications, books, and online recordings. These participants are added to a 6-month waitlist for a Cambridge Health Alliance mindfulness-based intervention group. All participants are scheduled to meet with their primary care provider during week 6 for a collaborative action planning visit.
  Other Names: 6-month waitlist
  Arms: Mindfulness Intro. +resources +waitlist

SUMMARY:
Specific aims for this pilot study are:

(Behavioral health outcomes aim): Among primary care patients, compare the effectiveness of an 8-week mindfulness-based intervention (Mindfulness Training for Primary Care[MTPC]) vs. a 60-minute introduction to mindfulness plus referral to community resources on measures related to anxiety, depression, and stress, and self-management of chronic illness.

(Medical Regimen Adherence Aim): Among primary care patients, compare the effectiveness of MTPC vs. 60-minute introduction to mindfulness on the initiation and maintenance of an action plan.

(Patient-Provider Relationship Aim): To examine the effects of level of primary care provider mindfulness training on successful referral to program, patient-provider relationship measures, and on patient action plan initiation and maintenance.

DETAILED DESCRIPTION:
This project aims evaluate the integration of mindfulness training into the heart of the standard healthcare delivery system.

The investigators and collaborators have developed an 8-week mindfulness-based intervention for primary care called Mindfulness Training for Primary Care (MTPC). MTPC combines common Mindfulness-Based Intervention skills with additional attention to patient/provider relationships, cultural and socio-economic diversity, coping with chronic illness, reducing unnecessary medical care, and encouraging self-management skills acquisition.

This project addresses important gaps in the current mindfulness research and delivery system by evaluating the integration of the novel MTPC model into a system of urban, community, multi-cultural, safety-net Patient-Centered Medical Homes.

In this pilot randomized controlled trial, the investigators compare the effectiveness of 8-week MTPC versus a 60-minute introduction to mindfulness plus referral to community mindfulness resources for primary care patients on behavioral health outcomes of anxiety, depression, stress, and self-management of chronic illness. The investigators are also testing the effect of MTPC on rates of initiation and maintenance of health action plans that patients collaborate on with their primary care provider during study Week 6 . This study also enrolls primary care providers who have participated in various levels of mindfulness training, i.e., 16-hour and 8-week mindfulness-based stress reduction and 10-month mindful communication vs. no training.

Outcome assessments are conducted at baseline and study week 8. An action-planning visit with PCPs occurs at week 6 with follow-up during week 8 (initiation) and interview at study week 24 (maintenance).

ELIGIBILITY:
Inclusion Criteria:

* Current CHA patient with an enrolled CHA primary care doctor.
* CHA patients 18 years of age and older.
* Able to tolerate and participate in interviews and engage in all procedures.
* Able to give written consent in English OR willing and able to provide consent and complete assessments through a professional language translator when necessary.
* Diagnosis eligible to be covered by insurance for group visits (e.g., anxiety disorder, depression, or adjustment disorder related to chronic illness, pain, etc.).

Exclusion Criteria:

* Any cognitive impairment that precludes informed consent.
* Patients who, in the opinion of the Principal Investigator, pose an imminent risk of suicide or danger to self or others.
* Likelihood of potential incarceration such as a conviction or pending charges that may potentially result in imprisonment.
* Previous enrollment or randomization of treatment in the present study within the 12 months.
* Behaviors that may cause disruption to a mindfulness group.
* Patients with symptoms of psychosis, thought disorder, and/or severe mental illness, including schizophrenia, schizoaffective, bipolar disorder, or a current severe episode of major depressive disorder.
* Lack of insurance coverage for group psychotherapy may preclude participation in groups.
* Patients in their third trimester of pregnancy who foresee conflicts that preclude their commitment to completing all activities.
* Patients with highly unstable medical problems that put them at a high risk of hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale | Week 8
  The Perceived Stress Scale (PSS) (10 items) measures the degree to which situations in life are stressful. Items are designed to evaluate how overloaded, unpredictable, and uncontrollable one finds one's life. Each item is scored on a 5 point Likert scale from 0 (Never) to 4 (Very often).
Change in Patient Reported Outcomes Measurement Information System - Anxiety Short Form (PROMIS-ASF) | Week 8
  The Patient Reported Outcomes Measurement Information System - Anxiety Short Form 8a (PROMIS-ASF) is an 8-item scale used to assess patient-reported health status for anxiety. PROMIS instruments are funded by the National Institutes of Health (NIH) and used to reliably and validly measure patient-reported outcomes for clinical research and practice. Participants are asked to rate their experience of the item in the past seven days on a 5-point scale from 1 (Never) to 5 (Always). Ratings from baseline will be compared to ratings from 8 Weeks post-baseline.
Change in Patient Reported Outcomes Measurement Information System - Depression Short Form (PROMIS-DSF) | Week 8
  The Patient Reported Outcomes Measurement Information System - Depression Short Form 8a (PROMIS-DSF) is an 8-item scale used to assess patient-reported health status for depression. PROMIS instruments are funded by the National Institutes of Health (NIH) and used to reliably and validly measure patient-reported outcomes for clinical research and practice. Participants are asked to rate their experience of the item in the past seven days on a 5-point scale from 1 (Never) to 5 (Always). Ratings from baseline will be compared to ratings from 8 Weeks post-baseline.
Change in Self-Efficacy for Managing Chronic Disease (SECD-6) | Week 8
  The Self-Efficacy for Managing Chronic Disease Scale (SECD-6) is a 6-item scale that is used to evaluate a participant's ability to self-manage care for a chronic disease. SECD-6 asks participants to rate their confidence in their own ability to do certain activities, on a scale from 1 (not at all confident) to 10 (totally confident).
Action Plan Initiation Survey (APIS-5) | Week 8
  Patient self-reported Action Plan Initiation Survey (APIS-5) will be administered at post-treatment (PT Study Week 8). This 5-item questionnaire is adapted from a measure used by Guck et al. In this questionnaire, patients are asked to list their action plan goals generated with their PCP, and determine whether they met or did not meet each goal. For each unmet goal, patients are asked to rate the cause of not meeting the goal on an attributional rating scale using a 7-point format.

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire (FFMQ) | Week 8
  The Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item scale that examines five factors that represent aspects of the current empirical conception of mindfulness. These five facets include: "observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience." Participants rate their degree of agreement with each of the items on a Likert-type scale ranging from 1 (Never or very rarely true) to 5 (Very often or always true), with higher scores indicating higher experience of mindfulness.
Self-Compassion Scale-Short Form (SCS-SF) | Week 8
  The short-form Self-Compassion Scale (SCS-SF) is an abbreviated 12-item form of the original 26-item Self-Compassion Scale. The scale is scored on a 5 point Likert scale (1 = Almost never; 5 = Almost always), and negative subscale items are reverse scored.
Difficulty in Emotion Regulation Scale (DERS) | Week 8
  The Difficulties in Emotion Regulation (DERS) Scale is a 36-item self-report scale designed to assess emotional dysregulation.
Multidimensional Assessment of Interoceptive Awareness (MAIA) | Week 8
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item self-report scale designed to assess multiple aspects of interoception and interoceptive awareness.
Perceived Control Questionnaire (PCQ) | Week 8
  The Perceived Control Questionnaire (PCQ) is adapted from a 5-item perceived control measure from Jerant et al. and a previously validated survey from Armitage et al. This 5-item scale asks participants to rate their sense of control over chronic illness self-management on a 7-point scale from 1 (None) to 7 (Total).
Patient Activation Measure (PAM) | Week 8
  The Patient Activation Measure (PAM) is a 13-item scale that is designed to evaluate a participant's ability to be an effective and informed manager of his or her own health and health care. Participants are asked to rate their agreement with each statement on a 0-100 metric where 0 = the lowest possible activation and 100 = the highest possible activation as measured by this set of items.

OTHER OUTCOMES:
Action Plan Assessment (APA-10) | Week 6
  Action Plan Assessment (APA-10) (10 items) - this is a questionnaire to be completed after the PCP Visit, at PT Study Week 6. This 10-item scale evaluates patient behavior in the domains of self-determination, motivation, shared decision-making, and barrier appraisal. Participants are asked to rate their agreement with a statement on a 7-point scale from 1 (Strongly Disagree) to 7 (Strongly Agree).
Action Plan Follow-Up Interviews | Week 24
  Action Plan Follow-Up Interviews will be conducted by a blinded member of the MINDFUL-PC study staff at Follow-Up (6-months post-baseline). This staff member will contact patients after 6 months to ask about the status of the specific primary behavior focused on in the action plan. Staff members will rate patient behavior on a scale from -1 (Behavior is worse than baseline) to 3 (Behavior has exceeded the original expectations and other health behaviors have also improved).

CONTACTS AND LOCATIONS:
Overall Officials: Zev D Schuman-Olivier, MD, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance Center for Mindfulness and Compassion, Somerville, Massachusetts, United States

REFERENCES:
- [Background] Mccubbin T, Dimidjian S, Kempe K, Glassey MS, Ross C, Beck A. Mindfulness-based stress reduction in an integrated care delivery system: one-year impacts on patient-centered outcomes and health care utilization. Perm J. 2014 Fall;18(4):4-9. doi: 10.7812/TPP/14-014. PMID 25662520
- [Background] Merkes M. Mindfulness-based stress reduction for people with chronic diseases. Aust J Prim Health. 2010;16(3):200-10. doi: 10.1071/PY09063. PMID 20815988
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Chiesa A, Serretti A. Mindfulness based cognitive therapy for psychiatric disorders: a systematic review and meta-analysis. Psychiatry Res. 2011 May 30;187(3):441-53. doi: 10.1016/j.psychres.2010.08.011. Epub 2010 Sep 16. PMID 20846726
- [Background] Holzel BK, Lazar SW, Gard T, Schuman-Olivier Z, Vago DR, Ott U. How Does Mindfulness Meditation Work? Proposing Mechanisms of Action From a Conceptual and Neural Perspective. Perspect Psychol Sci. 2011 Nov;6(6):537-59. doi: 10.1177/1745691611419671. PMID 26168376
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Schuman-Olivier Z, Hoeppner BB, Evins AE, Brewer JA. Finding the right match: mindfulness training may potentiate the therapeutic effect of nonjudgment of inner experience on smoking cessation. Subst Use Misuse. 2014 Apr;49(5):586-94. doi: 10.3109/10826084.2014.850254. PMID 24611853
- [Background] Alegria M, Sribney W, Perez D, Laderman M, Keefe K. The role of patient activation on patient-provider communication and quality of care for US and foreign born Latino patients. J Gen Intern Med. 2009 Nov;24 Suppl 3(Suppl 3):534-41. doi: 10.1007/s11606-009-1074-x. PMID 19842003
- [Background] Neff KD, Germer CK. A pilot study and randomized controlled trial of the mindful self-compassion program. J Clin Psychol. 2013 Jan;69(1):28-44. doi: 10.1002/jclp.21923. Epub 2012 Oct 15. PMID 23070875
- [Background] Wiegner L, Hange D, Bjorkelund C, Ahlborg G Jr. Prevalence of perceived stress and associations to symptoms of exhaustion, depression and anxiety in a working age population seeking primary care--an observational study. BMC Fam Pract. 2015 Mar 19;16:38. doi: 10.1186/s12875-015-0252-7. PMID 25880219
- [Background] Benzo RP. Mindfulness and motivational interviewing: two candidate methods for promoting self-management. Chron Respir Dis. 2013 Aug;10(3):175-82. doi: 10.1177/1479972313497372. PMID 23897933